CLINICAL TRIAL: NCT03675841
Title: A Phase I，Pazufloxacin Mesilate Ear Drops in Patients With Chronic Suppurative Otitis Media
Brief Title: Pazufloxacin Mesilate Ear Drops in Patients With Chronic Suppurative Otitis Media
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZK-PZFX-201704
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Chronic Suppurative Otitis Media
Keywords: Pazufloxacin Mesilate ear drops
MeSH Terms: interventions — Urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.1% single-dose pre (Experimental): Three subjects will be treated with Pazufloxacin Mesilate ear drops 0.1% single dose
  Interventions: Drug: Pazufloxacin Mesilate ear drops
- 0.1% single-dose (Experimental): Ten subjects will be treated with Pazufloxacin Mesilate ear drops 0.1% single dose
  Interventions: Drug: Pazufloxacin Mesilate ear drops
- 0.3% single-dose (Experimental): Ten subjects will be treated with Pazufloxacin Mesilate ear drops 0.3% single dose
  Interventions: Drug: Pazufloxacin Mesilate ear drops
- 0.5% single-dose (Experimental): Ten subjects will be treated with Pazufloxacin Mesilate ear drops 0.5% single dose
  Interventions: Drug: Pazufloxacin Mesilate ear drops

INTERVENTIONS:
Drug: Pazufloxacin Mesilate ear drops — Pazufloxacin Mesilate ear drops of 0.1%，0.3%，0.5%
  Other Names: ear drops

SUMMARY:
Objective To observe the safety and tolerability of Pazufloxacin Mesylate Ear Drops of different concentrations in patients with simple chronic suppurative otitis media.

DETAILED DESCRIPTION:
The test group was completed in sequence from low to high concentrations, and safety tolerance was assessed after administration in one concentration group to determine whether to conduct follow-up group studies and, if necessary, adjust sampling time points according to pre-experimental results.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18-65 years old. Men and women are not restricted.
2. Clinical diagnosis of simple chronic suppurative otitis media with ear effusion secretion, tympanic membrane perforation about 2 mm, the need for local use of antibiotics in patients.
3. Voluntarily sign written informed consent.
4. Non-breast-feeding women volunteered to take appropriate contraceptive measures (including abstinence, intrauterine devices, diaphragms and spermicides) during the study period (screening period to one week after administration). Men are willing to use approved contraceptive methods (including the use of condoms and spermicides or the use of oral, implantable or injectable contraceptives by their partners, intrauterine devices, diaphragms and spermicides) or sexual partner infertility.

Exclusion Criteria:

1. Quinolone antibiotics allergy and severe allergic constitution.
2. During the study, ear fluid could not be collected.
3. Patients with severe need for systemic use of antibiotics.
4. Infections caused by pathogens such as fungi and viruses (bullous tympanitis).
5. Patients with cholesteatoma.
6. Complicated with symptoms of extraaural infection (such as periaural cellulitis, mumps) or intracranial and extracranial complications (such as meningitis, brain abscess, thrombophlebitis of sigmoid sinus, subperiosteal abscess of the ear, Bezold's abscess of the neck).
7. Suffer from severe brain, heart, lung, liver, kidney and blood diseases.
8. People suffering from severe diseases that affect their survival, such as malignant tumors or AIDS, etc.
9. Abnormal liver and kidney function (ALT, Angiotensin sensitivity test(AST) ≥ 1.5 times the upper limit of normal value), creatinine clearance rate < 60ml/min).
10. Use any local or systemic antibiotics in the first 3 days of the admission.
11. Use any quinolones within the first 7 days of admission.
12. There were smokers who smoked more than 5 cigarettes a day within one year.
13. There was a history of alcoholism and drug abuse within one year.
14. Diagnosis of diabetes or poor blood glucose control.
15. Those who are unable to cooperate or unwilling to cooperate with neuropsychiatric disorders.
16. Pregnant or lactating women, those who do not use contraceptive measures as required, or those who are unwilling to take contraceptive measures.
17. Patients who took part in other clinical trials in the first 3 months.
18. Blood donation within three months before admission, or intended during or three months after the end of the trial or blood components.
19. Researchers believe that patients who are not fit to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-07-29 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-06-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Within two days after administration
  Objective To observe the safety and tolerability of Pazufloxacin Mesylate Ear Drops of different concentrations in patients with simple chronic suppurative otitis media.

SECONDARY OUTCOMES:
Cmax | Within two days after administration
  Pharmacokinetics
Tmax | Within two days after administration
  Pharmacokinetics
Area under concentration time curve | Within two days after administration
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: lei chen, PHD, Study Director — Jiangsu Province People's Hospital
Locations (1):
- Jiangsu Province People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No